CLINICAL TRIAL: NCT01385683
Title: Investigation Drug-drug Interaction Between Dabigatran and Clarithromycin
Acronym: IMAGINE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Groupe de Recherche sur la Thrombose (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 1008073; 2010-024047-33 (EudraCT Number)
Record Dates: First submitted 2011-06-27; First posted 2011-06-30 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: Healthy volunteer; Pharmacokinetic; pharmacodynamic; Polymorphism, Genetic
MeSH Terms: interventions — Clarithromycin; Dabigatran

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Dabigatran then dabigatran and clarithromycin
  Interventions: Drug: Dabigatran then dabigatran and clarithromycin
- Arm B (Active Comparator): Clarithromycin and dabigatran and dabigatran
  Interventions: Drug: Clarithromycin and dabigatran then dabigatran

INTERVENTIONS:
Drug: Dabigatran then dabigatran and clarithromycin — D4 : dabigatran 300 mg (4 tablets) one time. D8 to D10 : Clarithromycin 500mg (1 tablet) twice daily. D11 : Clarithromycin 500mg (1 tablet) + 300mg dabigatran (4 tablets)
  Other Names: Dabigatran (Pradaxa)75 mg; Clarithromycin (Zeclar) 500 mg
  Arms: Arm A
Drug: Clarithromycin and dabigatran then dabigatran — D1 to D3 : Clarithromycin 500mg (1 tablet) twice daily. D4 : Clarithromycin 500mg (1 tablet) + 300mg dabigatran (4 tablets). D11 : dabigatran 300 mg (4 tablets) one time.
  Other Names: Dabigatran (Pradaxa) 75 mg; Clarithromycin (Zeclar) 500 mg
  Arms: Arm B

SUMMARY:
Dabigatran (Pradaxa ®) is a new oral anticoagulant. It is used to prevent venous thromboembolism in orthopedic surgery and has recently demonstrated efficacy and safety at least as good as anticoagulants in the prevention of thromboembolism in atrial fibrillation and the treatment of venous thromboembolism. It is administered with fixed dose and does not require laboratory monitoring because of the low inter and intra individual pharmacokinetic (PK) and pharmacodynamics (PD) of dabigatran. However, the bioavailability of dabigatran is very low (6.5%) and is controlled by an efflux protein, P-GP. This molecule has a genetic polymorphism. The inhibition of this protein can cause a significant increase in intestinal absorption of dabigatran and expose patients to a risk of bleeding by overdose. Two major drug interactions have been identified : quinidine (cons-indication) and amiodarone (precautions). It is likely that other interactions exist and can be clinically significant in patients not selected such as testing. The development of tools to study the influence of P-GP on the PK and PD of dabigatran is therefore interesting. As the P-GP has a genetic polymorphism, the study of the latter is an important element in the detection of drug interactions. In this sense, clarithromycin, a potent inhibitor of P-GP is a good model to evaluate the primary mechanism of drug interaction of dabigatran and optimize the experimental design of studies to be conducted.

ELIGIBILITY:
Inclusion Criteria:

* affiliated or beneficiary of a social security category
* having signed the inform consent form
* having signed the genetic consent form
* weight between 60 and 85 kg
* normal clinical exam
* normal biological exam

Exclusion Criteria:

* contra-indication to dabigatran
* contra-indication to clarithromycin
* previous history of psychiatric disease, or antidepressant treatment, or convulsion, or hemorrhagic disease
* smoker
* peptic ulcer
* severe liver disease
* severe kidney failure
* previous surgery within one month

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Determination of dabigatran and its metabolites in plasma by LC/MS-MS method | At Day 4 and Day 11
  Calculating the area under the curve (AUC) from plasma concentrations of dabigatran versus time by the trapezoidal method. Determination of maximum concentration (Cmax)

SECONDARY OUTCOMES:
Pharmacodynamic parameters | At Day 4 and Day 11
  Measures activated Partial Thromboplastin Time (aPTT)and measures ECarin Time (ECT),
Genotyping | At Day 1
  Genotyping of MDR-1 (gene for P-GP): C3435T SNP of exon 26, SNP G2677T / A of exon 21 and C1236T SNP of exon 12

CONTACTS AND LOCATIONS:
Overall Officials: Patrick MISMETTI, MD PhD, Principal Investigator — CHU de Saint-Etienne; Xavier DELAVENNE, Pharmacist, Study Chair — CHU de Saint-Etienne
Locations (1):
- Service de Medecine et Therapeutique, Saint-Etienne, France